CLINICAL TRIAL: NCT05120024
Title: Multicenter Non-interventional Retro- and Prospective Safety and Efficacy Study of Prolgolimab (Forteca - Anti-PD1) in Patients With Advanced Melanoma (FOrteca Real Practice Assessment)
Brief Title: Multicenter Study of Safety and Efficacy of Prolgolimab in Patients With Advanced Melanoma in Routine Clinical Practice
Acronym: FORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MelanomaPRO, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: FORA
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describe the safety, tolerability, efficacy and approaches to prescribing prolgolimab in the standard dosing regimen of 1 mg / kg every 2 weeks in patients with advanced melanoma in routine practice.

Prolgolimab (Forteca, formerly BCD 100) is an IgG1 anti-PD-1 (programmed cell death protein 1) monoclonal antibody containing the Fc-silencing 'LALA' mutation.

DETAILED DESCRIPTION:
Describe the safety and tolerability of using Prolgolimab at a standard dosage regimen of 1 mg / kg every 2 weeks.

Describe the efficacy of prolgolimab 1 mg / kg every 2 weeks in patients with metastatic or inoperable melanoma in routine practice, based on the following indicators: Progression-free survival (time from first dose of prolgolimab to disease progression or death for any reason); Overall survival (time from receiving the first dose of prolgolimab to death for any reason); Objective response rate (proportion of patients with a complete or partial response to prolgolimab therapy).

ELIGIBILITY:
Inclusion Criteria:

Histological confirmed melanoma Advanced stage (unresectable III or metastatic IV) Treated by at least one therapy line including prolgolimab in routine practice -

Exclusion Criteria:

- Patient participation in any interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced melanoma, who were treated by prolgolimab (anti-PD1) in routine clinical practice in Russian Federation
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events during prolgolimab therapy | 2 years
  The rate of all grade and grade 3-5 adverse events and the rate of discontinuation of study drug(s) due to adverse events.
Objective response rate | 3 years
  The response rate during prolgolimab therapy in patients with unresectable advanced melanoma

SECONDARY OUTCOMES:
Progression free survival (PFS) | 3 years
  The median PFS and 24 months PFS rate of patients with advanced melanoma during prolgolimab
Overall survival (OS) | 3 years
  The median OS and 24 months OS rate of patients with advanced melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Orlova, MD PhD, Study Chair — MelanomaPRO, Russia
Locations (1):
- N.N. Blokhin National Medical Research Center of Oncology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided